CLINICAL TRIAL: NCT04065919
Title: Evaluation of Liposomal Bupivacaine Compared to Usual Care and Its Effects on Pain for Cardiac Surgery
Acronym: EXPAREL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Florida Heart and Lung Institute (Other)
Responsible Party: Principal Investigator, Charles Klodell, MD, Cardiothoracic Surgeon, Florida Heart and Lung Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIT#2018-137
Record Dates: First submitted 2019-08-02; First posted 2019-08-22 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Cardiothoracic Surgery
MeSH Terms: interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Intervention Model Description: Study comparing current standard of therapy using 0.25% bupivacaine with epinepherine at 1cc/kg total dose and the addition of liposomal bupivacaine 266mg/20ml for pain management in cardiac surgery. Patient and Investigator are blinded.
Who Masked: Participant, Investigator
Masking Description: Patients will be randomized per study coordinator. SOC includes 0.25%bupivacaine with epinephrine at 1cc/kg total dose and the treatment arm will include liposomal bupivacaine 266mg/20ml added to usual dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exparel (Active Comparator): administration of liposomal bupivacaine 266mg/20mL+ 40 mL bupivacaine 0.25% bupivacaine
  .
  Interventions: Drug: Liposomal bupivacaine; Drug: 0.25% Bupivacaine with epinephrine
- Standard of Therapy (Active Comparator): administration of 0.25% bupivacaine with epinephrine at 1cc/kg total dose
  Interventions: Drug: 0.25% Bupivacaine with epinephrine

INTERVENTIONS:
Drug: Liposomal bupivacaine — 20mL EXPAREL+40mL bupivacaine 0.25% infiltrated into 5th intercostal space
  Other Names: Exparel
  Arms: Exparel
Drug: 0.25% Bupivacaine with epinephrine — 0.25% Bupivacaine with epinephrine at 1cc/kg total dose infiltrated into 5th intercostal space

SUMMARY:
Evaluation of Liposomal Bupivacaine Compared to Usual Care and its Effect on Pain for Cardiac Surgery

DETAILED DESCRIPTION:
Current standard of care for pain management includes a multimodal approach of peristernal and fifth intercoastal infiltration with 0.25% bupivacaine with epinepherine combined with immediate post operative IV acetaminophen, followed by scheduled oral acetaminophen and supplemental IV and PO narcotics. This practice is beneficial since it controls most of the direct surgical site pain for at least 6 hours, however, after the local anesthetic dissipates, pain is usually managed with the use of opioids combined with scheduled oral acetaminophen.

Opioids are the most commonly used medications to control pain early after surgery because of their high potency. However, their undesirable effects and risk of dependence become limitations.

The Investigators believe Liposomal Bupivacaine would be beneficial in this population due to its quick onset of action and prolonged half-life associated with liposomal formulation ranging from 23.8 to 34.1 hours. The primary endpoint will be a 20% reduction in opioids use.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* All open heart surgeries from September 1, 2019 - September 30, 2020
* Able to read, comprehend and sign the informed consent form

Exclusion Criteria:

* Pregnancy
* < 18 years old and prisoners
* Not able to sign informed consent, including patients with an (LAR) legally authorized representative
* Patients with chronic pain requiring scheduled narcotic use
* Stage 4 kidney disease, Child Pugh score suggestive of liver cirrhosis/ disease
* Recent MI within 7 days of scheduled Cardiac surgery
* Known allergy to Liposomal Bupivacaine or derivative of
* Have or is currently involved in a Research Study within 30 days of scheduled surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
20% change in opioids use | From post operative day of cardiac surgery through length of hospital admission and through study completion, an average of one year.
  Record daily narcotic use

SECONDARY OUTCOMES:
Time to extubation | Post operative day of surgery through study completion, an average of 1 year
  Record in 15 minutes intervals the time when the breathing tube is removed
Time to ICU | Post operative day of surgery through study completion, an average of 1 year
  Record time in 15 minute intervals the length of time in ICU
Pain Scores on Post op day 2,3 and 4 | Post operative day of cardiac surgery through Post operative Day 4
  Record pain scores using the Wong - Baker" FACES" Pain rating scale and /or CPOT Critical Care Pain Observation Tool. Collecting the Scale ratings of 4-10.*Face #4 Hurts a Little, Face#6 Hurts Even More, Face #8 Hurts a Whole Lot Face#10 Hurts Worst. CPOT- Critical Care Pain Observational Tool Documenting Pain Intensity, Pain Location, Pain Radiation and Pain Description.
Total narcotic use on Post op Day 2,3, and 4 | Day of cardiac surgery to Post op day 4
  Record daily narcotic use both Oral and Intravenous administration
Time to Hospital Discharge | Count the number of days from admission for cardiac surgery to day of hospital discharge through study completion , an average of one year
  Record the number of days(LOS) length of stay in the hospital from post operative surgery to discharge
Major Adverse Cardiac Effects of Liposomal Bupivacaine | Time of peristernal and fifth intercostal infiltration of liposomal bupivacaine through the expected half life associated with liposomal formulation ranging from 23.8 up to 34.1 hours.
  Record Major Adverse Cardiac Effects associated with Liposomal Bupivacaine, Arrythmias, Hypotension > 90/50,AV Block and Cardiac Arrest

CONTACTS AND LOCATIONS:
Overall Officials: Charles T Klodell, MD, Principal Investigator — Florida Heart and Lung Institute, HCA Physician Services
Locations (1):
- Florida Heart and Lung Institute, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No